CLINICAL TRIAL: NCT07405944
Title: Vericiguat's Effects on Reverse Remodeling Indices: Pathophysiologic Approach to Treatment of Heart Failure With Reduced Ejection Fraction
Brief Title: Vericiguat and Reverse Remodeling Indices in Heart Failure
Acronym: VERI-PATH
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Collaborators: Slovenian Research Agency (Other)
Responsible Party: Principal Investigator, Gregor Poglajen, Associate Professor, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0120-5/2025-2711-3
Record Dates: First submitted 2025-11-22; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Heart Failure With Reduced Ejection Fraction (HFrEF); Chronic Heart Failure
Keywords: Vericiguat; Soluble Guanylate Cyclase; Cyclic GMP; Reverse Remodeling; Cardiac Magnetic Resonance Imaging; Myocardial Perfusion Imaging; Fibrosis; Inflammation; Angiogenesis; Oxidative Stress; Immunomodulation; Insulin Resistance
MeSH Terms: conditions — Fibrosis; Inflammation; Insulin Resistance | interventions — vericiguat

STUDY DESIGN:
Intervention Model Description: Two-arm randomized (1:1), parallel assignment of vericiguat plus guideline-directed medical therapy versus usual care alone for 12 months. Non-randomized open-label extension for prior control participants in Months 12-24 (exploratory).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vericiguat + GDMT (Experimental): Participants will receive vericiguat added to guideline-directed medical therapy (GDMT) for heart failure. Vericiguat will be initiated at 2.5 mg once daily and up-titrated in approximately 2-week intervals to 5 mg and then a target dose of 10 mg once daily, as tolerated, over the 12-month randomized phase.
  Interventions: Drug: Vericiguat; Drug: Guideline Directed Medical Therapy for Heart Failure (GDMT)
- GDMT (Active Comparator): Participants will continue to receive guideline-directed medical therapy (GDMT) for heart failure without vericiguat during the 12-month randomized phase (vericiguat offered during exploratory extension).
  Interventions: Drug: Guideline Directed Medical Therapy for Heart Failure (GDMT)

INTERVENTIONS:
Drug: Vericiguat — Oral soluble guanylate cyclase stimulator administered once daily, initiated at 2.5 mg and up-titrated in approximately 2-week intervals to 5 mg and then 10 mg as tolerated, in addition to guideline-directed medical therapy for heart failure.
  Other Names: Verquvo; MK-1242
  Arms: Vericiguat + GDMT
Drug: Guideline Directed Medical Therapy for Heart Failure (GDMT) — Standard combination heart failure therapy according to current guidelines (ARNI, beta-blocker, MRA, and SGLT2 inhibitor as tolerated).
  Other Names: GDMT

SUMMARY:
The goal of this clinical trial is to investigate how vericiguat benefits adults with stable heart failure with reduced ejection fraction (HFrEF) who are already receiving guideline-directed medical therapy.

The main questions are:

* Does vericiguat improve right ventricular systolic function, measured by tricuspid annular plane systolic excursion (TAPSE)?
* Does vericiguat favourably influence myocardial remodeling, fibrosis, angiogenesis, inflammation, metabolism, renal function, and hematologic balance?
* Do genetic and oxidative stress profiles modify treatment response? Researchers will compare a group receiving vericiguat plus usual care with a group receiving usual care alone to assess structural, functional, and biomarker changes over 12 months.

Participants will:

* Have blood drawn at baseline and follow-up visits for biomarker, metabolomic, genetic, transcriptomic, and hematologic analyses, including platelet function testing
* Perform oral glucose tolerance tests (OGTT) to assess insulin resistance
* Undergo echocardiography, cardiac magnetic resonance imaging, and cardiac scintigraphy to evaluate heart structure, function, and perfusion
* Attend follow-up visits at 1, 3, 6, and 12 months Open-label extension: After the 12-month randomized phase, participants originally assigned to usual care will be offered open-label vericiguat and followed for an additional 12 months. This exploratory extension will reassess study outcomes to evaluate the consistency and magnitude of response to vericiguat in the prior control cohort.

DETAILED DESCRIPTION:
Heart failure with reduced ejection fraction (HFrEF) involves pathologic processes that lead to maladaptive remodeling of the myocardium with ventricular dilation, wall thickening, and cellular and microvascular changes that progressively worsen cardiac function. Many established therapies for heart failure can promote reverse remodeling, improving symptoms and long-term outcomes.

Vericiguat is a soluble guanylate cyclase (sGC) stimulator that increases cyclic guanosine monophosphate (cGMP), a signaling molecule with vasodilatory and cardioprotective effects that is impaired in heart failure. Randomized trials show that vericiguat reduces the risk of worsening heart-failure events in HFrEF after recent decompensation, and emerging evidence indicates that these benefits extend to stable HFrEF. The mechanisms by which vericiguat may benefit patients with HFrEF remain incompletely understood.

Preclinical data suggest that augmenting cGMP signaling may confer antifibrotic, antihypertrophic, antiinflammatory, proangiogenic, and metabolic effects. These mechanisms could contribute to reverse remodeling and improved clinical status, but they require confirmation in a clinical setting.

This randomized, controlled study will evaluate the effects of vericiguat on right ventricular systolic function, assessed by tricuspid annular plane systolic excursion (TAPSE), and will characterize associated structural and biologic changes in adults with stable HFrEF on contemporary GDMT. Sixty participants will be randomized to vericiguat plus usual care or to usual care alone and followed for 12 months, with study visits at 1, 3, 6, and 12 months.

At each visit, blood samples will be collected for analysis of circulating biomarkers reflecting fibrosis, inflammation, angiogenesis, renal function, and metabolism, as well as transcriptomic profiling. Comprehensive metabolomic profiling will be performed, and insulin resistance will be evaluated by oral glucose tolerance testing (OGTT) at baseline and 12 months. Hematologic parameters will be measured at each visit, while platelet function will be assessed at baseline and 12 months.

Cardiac structure and function will be assessed using transthoracic echocardiography, cardiac magnetic resonance imaging, and cardiac scintigraphy. Imaging will quantify biventricular volumes, systolic function, fibrosis, and perfusion.

The study will investigate whether cumulative oxidative stress and genetic variation modify the response to vericiguat. Cumulative oxidative stress will be quantified from serial 8-hydroxy-2'-deoxyguanosine (8-OHdG) measurements (area under the curve) and examined for interaction with treatment effects on TAPSE and other outcomes. Genetic analyses will assess variants in drug-disposition and NO-sGC-cGMP pathway genes for associations with response.

After completing the 12-month randomized phase, participants originally assigned to usual care will be offered open-label vericiguat and followed for an additional 12 months. This non-randomized, exploratory extension will re-measure the randomized-phase outcomes to evaluate the consistency and magnitude of response to vericiguat in the prior control cohort, using Month 12 values as the extension baseline.

Overall, this research is designed to clarify the pathophysiologic mechanisms of vericiguat therapy in HFrEF and to support more personalized treatment strategies for patients living with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from an adult patient (≥ 18 years old) to participate in the clinical study,
* Stable HFrEF defined as no heart failure worsening in the 6 months before randomization that required hospitalization or outpatient diuretic treatment,
* Confirmed diagnosis of chronic heart failure with reduced ejection fraction (LVEF ≤ 40%, confirmed by echocardiography) within 12 months before randomization,
* Stable GDMT for HFrEF for at least 3 months prior to randomisation.

Exclusion Criteria:

* Systolic blood pressure < 100 mmHg or symptomatic hypotension,
* Current or planned use of long-acting nitrates, soluble guanylate cyclase stimulators, or phosphodiesterase type V inhibitors,
* Known allergy/hypersensitivity to soluble guanylate cyclase stimulators,
* Awaiting heart transplantation or dependence on continuous inotropic therapy
* Cardiac amyloidosis, sarcoidosis, myocarditis, stress cardiomyopathy, or tachycardic cardiomyopathy,
* Acute coronary syndrome, coronary artery bypass grafting, or percutaneous coronary intervention in the past three months before randomisation,
* Long-term mechanical circulatory support of the left ventricle,
* Active infection,
* Chronic kidney disease stage 4 or 5, and
* Advanced liver failure classified as Child-Pugh B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in right ventricular systolic function assessed by right ventricular fractional area change (RV FAC) | Baseline to 6 months and 12 months
  Change in RV FAC (%), measured by transthoracic echocardiography (TTE) in the apical four-chamber view.

SECONDARY OUTCOMES:
Change in left ventricular systolic function assessed by left ventricular ejection fraction (LVEF) | Baseline to 6 months and 12 months
  Change in LVEF (%), measured by transthoracic echocardiography using 2D biplane Simpson's method.
Change in left ventricular systolic function assessed by left ventricular global longitudinal strain (GLS) | Baseline to 6 months and 12 months
  Change in left ventricular GLS (%), measured by transthoracic echocardiography using speckle-tracking.
Change in left ventricular structure assessed by left ventricular mass index (LVMI) | Baseline to 6 months and 12 months
  Change in LVMI (g/m²), calculated from transthoracic echocardiography using the Devereux formula and indexed to body surface area.
Change in right ventricular systolic function assessed by tricuspid annular plane systolic excursion (TAPSE) | Baseline to 6 months and 12 months
  Change in TAPSE (mm), measured by transthoracic echocardiography in the apical four-chamber view using M-mode.
Change in circulating serum fibrosis biomarkers assessed by Galectin-3 (Gal-3) and soluble ST2 (sST2) | Baseline, 1 month, 3 months, 6 months, and 12 months
  Change in serum Gal-3 (ng/mL) and sST2 (ng/mL) concentrations, measured in peripheral blood samples.
Change in serum angiogenetic biomarkers assessed by angiogenesis-related biomarker panel composite score | Baseline, 1 month, 3 months, 6 months, and 12 months
  Change in angiogenesis-related biomarker panel composite score, measured using a Luminex multiplex immunoassay (Human XL Cytokine Luminex® Performance Assay 46-plex).
Change in systemic inflammation assessed by serum inflammatory biomarker panel composite score | Baseline, 1 month, 3 months, 6 months, and 12 months
  Change in serum inflammatory biomarker panel composite score, measured using a Luminex multiplex immunoassay (Human XL Cytokine Luminex® Performance Assay 46-plex).
Change in cardiac fibrosis assessed by the extent of late gadolinium enhancement (LGE) | Baseline to 12 months
  Change in extent of myocardial LGE (% of left ventricular mass), quantified by cardiac magnetic resonance (CMR).
Change in myocardial microvascular dysfunction assessed by quantitative myocardial perfusion scintigraphy | Baseline to 12 months
  Change in myocardial blood flow (MBF, mL/min/g), measured by quantitative myocardial perfusion scintigraphy.
Change in insulin sensitivity assessed by the Matsuda index | Baseline and 12 months
  Change in insulin sensitivity measured by the Matsuda index (unitless), derived from a standard 75-g oral glucose tolerance test (OGTT).
Change in kidney function assessed by urine albumin-to-creatinine ratio (UACR) | Baseline, 1 month, 3 months, 6 months, and 12 months
  Change in UACR (mg/g), measured from a spot urine sample.

OTHER OUTCOMES:
Difference in right ventricular systolic function assessed by right ventricular fractional area change (RV FAC) between genotype groups | Genotyping at baseline; RV FAC change from baseline to 12 months
  Difference in change in RV FAC (%), measured by transthoracic echocardiography, between patients with wild-type vs mutated UGT1A9 gene, assessed by genotyping/sequencing from peripheral blood samples.
Change in pre-specified gene set expression score, assessed by peripheral blood RNA-seq | Baseline, 1 month, 3 months, 6 months, and 12 months
  Change in expression score of a pre-specified gene set (unitless normalized RNA-seq expression score), assessed by peripheral blood RNA sequencing (RNA-seq).
Difference in right ventricular systolic function assessed by right ventricular fractional area change (RV FAC) between high versus low oxidative stress groups | Time Frame: 8-OHdG at baseline, 1 month, 3 months, 6 months, and 12 months; RV FAC change from baseline to 12 months
  Difference in change in RV FAC (%), measured by transthoracic echocardiography, between participants with high versus low oxidative stress defined by the median of the 12-month urinary 8-hydroxy-2'-deoxyguanosine (8-OHdG) area-under-the-curve (AUC, ng/mL·month), measured by validated immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Poglajen, MD, PhD, Principal Investigator — Advanced Heart Failure and Transplantation Center, Department of Cardiology, University Medical Centre Ljubljana, Ljubljana, Slovenia
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) that underlie the results reported in future publications (text, tables, figures, and appendices) will be shared upon reasonable request. Shared IPD will include baseline characteristics, outcome measures, and relevant biomarker data, excluding data that could compromise participant privacy or institutional confidentiality.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be made available within 6 months after publication of the main results and will remain accessible for at least 5 years thereafter.
Access Criteria: Researchers whose proposed use of the data is approved by the principal investigator will be granted access. Proposals should include a concise research plan and statistical analysis outline. Requests should be submitted to tine.bajec@kclj.si. Approved requesters will sign a data sharing agreement to ensure data confidentiality and appropriate use.